CLINICAL TRIAL: NCT04169802
Title: An Observational, Non-Significant Risk Study Of The Retinal Health Monitoring System (RHMS) - Visual Acuity Module - In Normal Patients And Patients With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Study Evaluating Retinal Health Monitoring System Visual Acuity Module.
Status: Completed | Type: Observational
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCT-201
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Age Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; visual acuity
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Normal subjects: Age ≥ 50 years, Corrected distance or near visual acuity (VA) of ≥ 20/25 Snellen equivalent, in the study eye.
  Interventions: Diagnostic Test: Retinal Health Monitoring System Visual Acuity Module; Diagnostic Test: Sloan letter, logarithmic near visual acuity chart (Reference Chart)
- Subjects with neovascular AMD: Age ≥ 50 years, History of neovascular age-related macular degeneration, in the study eye, Corrected distance or near VA of ≥ 20/200 Snellen equivalent, in the study eye.
  Interventions: Diagnostic Test: Retinal Health Monitoring System Visual Acuity Module; Diagnostic Test: Sloan letter, logarithmic near visual acuity chart (Reference Chart)

INTERVENTIONS:
Diagnostic Test: Retinal Health Monitoring System Visual Acuity Module — Assessment of corrected near visual acuity
Diagnostic Test: Sloan letter, logarithmic near visual acuity chart (Reference Chart) — Assessment of corrected near visual acuity

SUMMARY:
Assess the performance and usability of the RHMS Visual Acuity Module.

DETAILED DESCRIPTION:
This 510(k)-enabling study is designed to assess the performance and usability of the RHMS Visual Acuity Module in normal patients and patients with neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 - Normal subjects

1. Age ≥ 50 years
2. Corrected distance or near visual acuity (VA) of ≥ 20/25 Snellen equivalent, in the study eye
3. Able to perform self-testing with the Visual Acuity Module of the RHMS after training
4. Able and willing to give informed consent

Cohort 2 - Subjects with neovascular AMD

1. Age ≥ 50 years
2. History of neovascular age-related macular degeneration, in the study eye
3. Corrected distance or near VA of ≥ 20/200 Snellen equivalent, in the study eye

Exclusion Criteria:

Cohort 1 - Normal subjects

1. History of ophthalmic disease resulting in decrease in visual acuity per the Investigator, in the study eye
2. Use of any investigational drug in the past 30 days, or investigational, interventional device in the past 60 days

Cohort 2 - Subjects with neovascular AMD

1. History of geographic atrophy or macular atrophy within the central 3 mm of the macula, in the study eye
2. History of macular hole in the study eye
3. Use of any investigational drug in the past 30 days, or investigational, interventional device in the past 60 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged ≥ 50 years, with a normal central macula or with neovascular AMD
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the repeatability of CNVA measured by the RHMS Visual Acuity Module and the Reference Chart | 1 day
  To determine the precision (repeatability and reproducibility) of corrected near visual acuity (CNVA) measured by the RHMS Visual Acuity Module and an in-clinic, near logarithmic Sloan Letter chart (Reference Chart).
Comparison of the reproducibility of CNVA measured by the RHMS Visual Acuity Module and the Reference Chart | 1 day
  To evaluate the agreement of CNVA measured by the RHMS Visual Acuity Module and the Reference Chart
Agreement of CNVA measured by the RHMS Visual Acuity Module and the Reference Chart | 1 day
  To evaluate the usability of the RHMS Visual Acuity Module

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gregory, MD, Study Director — Kubota Vision Inc.
Locations (1):
- Retina Consultants of Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided